CLINICAL TRIAL: NCT01562795
Title: Efficacy of Nonsteroidal Anti-inflammatory Drugs in Treatment of Moderate and Severe Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangtian Zhou, MD, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xzhou
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Moderate to Severe Dry Eye Syndrome
MeSH Terms: interventions — Adrenal Cortex Hormones; Fluorometholone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group 1 (Experimental)
  Interventions: Drug: nonsteroid anti-inflammatory drops
- group 2 (Experimental)
  Interventions: Drug: nonsteroid anti-inflammatory drops
- group 3 (Experimental)
  Interventions: Drug: corticosteroids
- group 4 (Other)
  Interventions: Drug: artificial tear substitute

INTERVENTIONS:
Drug: nonsteroid anti-inflammatory drops — nonsteroid anti-inflammatory drops plus artificial tear substitute
  Other Names: prunoprefen
  Arms: group 1
Drug: nonsteroid anti-inflammatory drops — nonsteroid anti-inflammatory drops plus artificial tear substitute
  Other Names: bronuck
  Arms: group 2
Drug: corticosteroids — corticosteroids plus artificial tear substitute
  Other Names: Fluorometholone
  Arms: group 3
Drug: artificial tear substitute — artificial tear substitute alone
  Arms: group 4

SUMMARY:
This clinical trial is to investigate whether nonsteroid anti-inflammatory drops have therapeutic effect on moderate to severe dry eye patients.And compare the efficacy of the two nonsteroid anti-inflammatory drops with topical corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe dry eye syndrome
* tear film breakup time >0 second and ≤5 seconds,or schirmer test(no anaesthesia)≥2mm/5min and ≤5mm/5min
* corneal staining≥3 scores

Exclusion Criteria:

* allergic to any composition of the drugs under experiment
* previous use of anti-inflammatory drugs or immunosuppressive agent
* viral,bacterial or fungal infection of the eye
* eyelid anomaly
* glaucoma or high IOP
* significant meibomian gland dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
tear osmolarity | Day 0, Day 14

SECONDARY OUTCOMES:
corneal staining | 0 day,7th day and 14th day after treatment
Schirmer test(without anaesthesia) | 0 day,7th day,14th day after treatment
tear film breakup time(TBUT) | 0 day,7th day and 14th day after treatment
meibomian gland function | 0 day,7th day and 14th day after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, MD,PhD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China